CLINICAL TRIAL: NCT03551600
Title: Splanchnic and Renal Tissue Oxygenation During Enteral Feedings in Neonates With Patent Ductus Arteriosus
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Intermountain Health Care, Inc. (Other)
Responsible Party: Principal Investigator, Mariana Baserga, Principal Investigator, University of Utah
Other Study IDs: 83943
Record Dates: First submitted 2018-05-29; First posted 2018-06-11 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Infant, Premature; Congenital Heart Disease; Patent Ductus Arteriosus; Necrotizing Enterocolitis
Keywords: Near-infrared spectroscopy (NIRS); renal oxygen saturations; splanchnic oxygen saturations
MeSH Terms: conditions — Premature Birth; Heart Defects, Congenital; Ductus Arteriosus, Patent; Enterocolitis, Necrotizing | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Preterm, no PDA: Babies </= 32 weeks gestation at birth with no symptoms of a patent ductus arteriosus (PDA) or echocardiogram confirmation of no PDA
  Near-infrared spectroscopy (NIRS) monitoring x 48 hours of splanchnic and cranial regions, minimum of 8 feedings need to be recorded
  Interventions: Procedure: Near-infrared spectroscopy (NIRS)
- Preterm, moderate to large PDA: Babies </= 32 weeks gestation at birth with confirmed moderate to large PDA on echocardiogram Near-infrared spectroscopy (NIRS) monitoring x 48 hours of splanchnic and cranial regions, minimum of 8 feedings need to be recorded
  Interventions: Procedure: Near-infrared spectroscopy (NIRS)
- >/= 34 wk infants, no CHD: Babies >/= to 34 weeks gestation at birth with no evidence of ductal dependent congenital heart disease (CHD)
  Near-infrared spectroscopy (NIRS) monitoring x 48 hours of splanchnic, renal and cranial regions, minimum of 8 feedings need to be recorded
  Interventions: Procedure: Near-infrared spectroscopy (NIRS)
- >/= 34 week infants, CHD: Babies >/= to 34 weeks gestation at birth with ductal dependent CHD
  Near-infrared spectroscopy (NIRS) monitoring x 48 hours of splanchnic, renal and cranial regions, minimum of 8 feedings need to be recorded
  Interventions: Procedure: Near-infrared spectroscopy (NIRS)

INTERVENTIONS:
Procedure: Near-infrared spectroscopy (NIRS) — NIRS analyzes regional oxygen saturations (rSO2)

SUMMARY:
Patent ductus arteriosus (PDA) is a common problem in the neonatal intensive care unit and can be secondary to prematurity or congenital heart disease (CHD). PDA is the most common cardiovascular abnormality in preterm infants, and is seen in 55% of infants born at 28 weeks, and 1000 grams or less. In addition to producing heart failure and prolonged respiratory distress or ventilator dependence, PDA has been implicated in development of broncho-pulmonary dysplasia, interventricular hemorrhage, cerebral ischemia, and necrotizing enterocolitis (NEC). In an Israeli population study 5.6% of all very low birth weight infants (VLBW) were diagnosed with NEC, and 9.4% of VLBW infants with PDA were found to have NEC. In a retrospective analysis of neonates with CHD exposed to Prostaglandin E found that the odds of developing NEC increased in infants with single ventricle physiology, especially hypoplastic left heart syndrome. The proposed pathophysiological explanation of NEC and PDA is a result of "diastolic steal" where blood flows in reverse from the mesenteric arteries back into the aorta leading to compromised diastolic blood flow and intestinal hypo-perfusion. Prior studies have demonstrated that infants with a hemodynamically significant PDA have decreased diastolic flow velocity of the mesenteric and renal arteries when measured by Doppler ultrasound, and an attenuated intestinal blood flow response to feedings in the post prandial period compared to infants without PDA. Near Infrared Spectroscopy (NIRS) has also been used to assess regional oxygen saturations (rSO2) in tissues such as the brain, kidney and mesentery in premature infants with PDA. These studies demonstrated lower baseline oxygenation of these tissues in infants with hemodynamically significant PDA. These prior NIRS studies evaluated babies with a median gestational age at the time of study of 10 days or less. It is unknown if this alteration in saturations will persist in extubated neonates with PDA at 12 or more days of life on full enteral feedings.

In the present study the investigators hypothesize that infants with a PDA, whether secondary to prematurity or ductal dependent CHD, will have decreased splanchnic and renal perfusion and rSO2 renal/splanchnic measurements will be decreased during times of increased metabolic demand such as enteral gavage feeding. To test this hypothesis the investigators have designed a prospective observational study utilizing NIRS to record regional saturations at baseline, during feedings, and after feedings for 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* PDA secondary to prematurity

  1. Premature infants of ≤ 32 weeks gestational age at birth
  2. Patent ductus arteriosus diagnosed via echocardiogram
  3. Feeding volume ≥ 70 ml/kg/day
  4. Stable Clinical Condition (no vasopressors, no clinical sepsis)
  5. Age ≥ 12 days of life

Control group

1. Premature infants of ≤ 32 weeks gestational age at birth
2. No PDA
3. Feeding volume ≥ 70 ml/kg/day
4. Stable Clinical Condition (no vasopressors, no clinical sepsis)
5. Age ≥ 12 days of life

PDA secondary to CHD and Prostaglandin E (PGE)

1. Infants of ≥ 32 weeks gestational age at birth
2. Ductal dependant congenital heart disease
3. PGE infusion
4. No prior cardiac surgery
5. Any bolus feedings 10 ml/kg/day or more
6. Stable Clinical Condition (no vasopressors, no clinical sepsis)
7. Age ≥ 12 days of life

Control Group

1. Infants of ≥ 32 weeks gestational age at birth
2. No know congenital heart defect including PDA.
3. No prior cardiac surgery
4. Feeding volume ≥ 1/2 of total fluid volume ~50- 70 ml/kg/day
5. Stable Clinical Condition (no vasopressors, no clinical sepsis)

Exclusion Criteria:

* Lack of parental consent
* Multiple congenital anomalies
* Unstable clinical condition
* Prior abdominal pathology (medical/surgical necrotizing enterocolitis within the last 14 days, gastroschisis, or other abdominal abnormality)

Ages: 12 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm, Late preterm, and term infants
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Baseline renal and splanchnic rSO2 measurements | 48 hours
  Compare the baseline renal and splanchnic rSO2 measurements between preterm, late preterm, and term infants with a patent ductus arteriosus to those infants without a patent ductus arteriosus

SECONDARY OUTCOMES:
Renal and splanchnic rSO2 measurements during feedings | 48 hours
  Compare the renal and splanchnic rSO2 measurements between preterm, late preterm, and term infants with a patent ductus arteriosus to those infants without a patent ductus arteriosus immediately before, during, and after feedings

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Baserga, MD, Principal Investigator — University of Utah
Locations (3):
- United States (3):
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Health, Salt Lake City, Utah
  - Primary Children's Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No